CLINICAL TRIAL: NCT06177145
Title: Evaluation of the Effect "HASCV-R" Health Programme on Health Promoting and Protective Behaviours of the Turkish-Greek Population Exchange Migrant Women: a Randomized Controlled Trial
Brief Title: "HASCV-R" Health Programme
Acronym: HASCV-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Mehmet KORKMAZ, Phd. Mehmet Korkmaz, Asist. Prof. Department of Nursing, Bozok University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 01/20
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-12

CONDITIONS: Health Behavior
Keywords: Health behaviors; health promotion; Exchange migrant women
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: double-blind randomised controlled pretest-posttest experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): This study was carried out with the immigrant women living in Akdağmadeni district of Yozgat province. Trainings and measurement tools in the HASCV-R programme was implemented in the training centres in the neighbourhoods where immigrant women lived with the support of Akdağmadeni Lausanne Immigrants Association.
  Interventions: Other: HASCV-R program
- control (No Intervention)

INTERVENTIONS:
Other: HASCV-R program — "Healthy nutrition, Active life, Ways to cope with Stress, Cancer and cancer screening, Vaccination - Reproductive health" Training programme
  Arms: experimental

SUMMARY:
The goal of this randomized controlled trial: is to determine the effect of " HASCV-R " health programme on the health promoting and protective behaviours of the Turkish-Greek Population Exchange migrant women. The main question it aims to answer are:

• Does the HASCV-R program, positively affect the health promoting and protective behaviours of Turkish-Greek Population Exchange migrant women? The health program was given to the migrant women in the experimental group in five sessions of 40 minutes each for five weeks. The program was implemented to 48 migrant women. After obtaining consent from immigrant men, Data were gathered with all participants at the available time and places. The data were collected from the control and experimental groups at two different times, prior to the program was implemented and 3 months after the program was implemented.

DETAILED DESCRIPTION:
Health protection is the regulation of the environment in which the person lives both physically and socially. Health promotion, on the other hand, is defined as achieving optimal health, improving health by focusing on some cognitive factors and achieving optimal physical and mental health. The good quality of life of individuals is directly related to having health-protective and health-promoting behaviours. In the literature, there are training programmes to improve women's health, but there are no health-promoting and health-protective training programmes.

With the Lausanne Peace Treaty signed between Greece and Turkey in 1923, most of the Turks in Greece and Greeks in Turkey were subjected to forced migration. Thousands of Turks who were sent to Turkey after this agreement were settled in different parts of the country. Akdağmadeni district of Yozgat province is among these regions. These people and subsequent generations who experienced forced migration are called " Turkish-Greek Population Exchange ". The lifestyle, eating habits and cultures of the immigrants differ from the local people. In the literature, there is no health programme that improves or protects the health of immigrants. The unique value of this study is that it will be carried out with women who are immigrants and that the programme includes health-promoting and protective behaviours.

This research was conducted in accordance with the principles of double-blind randomised controlled pretest-posttest experimental research. In this research, the immigrant women do not know whether they are in the experimental or control group. The statistician conducting the research does not know which data belong to which group. In this way, blinding was done.

This study was carried out with the immigrant women living in Akdağmadeni district of Yozgat province. Trainings and measurement tools in the HASCV-R programme was implemented in the training centres in the neighbourhoods where immigrant women lived with the support of Akdağmadeni Lausanne Immigrants Association. The research was conducted between 15 May 2023 and 15 November 2023.

The population of the research consists of married women registered to Akdağmadeni Lausanne Mübadilleri Association residing in Akdağmadeni district centre where the research was conducted. The research was carried out with 2 different groups, 1 experimental group and 1 control group. According to the power analysis performed with G Power Clinic Calc programme, 45 experimental and 45 control groups were determined for 90% power and 0.05 type error. Considering the possibility of losses, the experimental group was increased by 10%. The study was planned to be carried out with 50 experimental and 50 control groups, with 5 substitutes for each group, totalling 100 married women who were immigrants. The study was conducted with 94 women, 48 experimental and 46 control groups.

Inclusion Criteria

* volunteering to participate in the study,
* be between the ages of 18 and 49,
* being a immigrant women,
* no communication barriers (to communicate with any problem such as hearing problem, speech impediment),
* to be married Exclusion Criteria
* being younger than 18 or over 49,
* be man,
* ınability to communicate with any problem such as hearing problem, speech impediment,
* living single,
* refusing to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study,
* be between the ages of 18 and 49,
* being a immigrant women,
* no communication barriers (to communicate with any problem such as hearing problem, speech impediment),
* to be married

Exclusion Criteria:

* being younger than 18 or over 49,
* be man,
* ınability to communicate with any problem such as hearing problem, speech impediment,
* living single,
* refusing to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire form | Prior to the program was implemented
  This form, developed by the researchers based on the literature, includes the socio-demographic characteristics of the men such as age, education status, income status, etc.).

SECONDARY OUTCOMES:
Health Promoting and Protective Behaviours Scale | prior to the program was implemented and 3 months after the program was implemented
  Evaluates the extent to which the individual keeps himself active in daily life, regular exercise behaviours and behaviours related to meeting physiological needs such as eating and drinking. Max:120, min;24
Scale for Determining Reproductive Health Protective Attitudes of Married Women | prior to the program was implemented and 3 months after the program was implemented
  It was developed to determine the reproductive health protective attitudes and behaviours of married women. Max; 50, min;10

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozturk, pHD, Principal Investigator — Bozok University
Locations (1):
- Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No